CLINICAL TRIAL: NCT05062746
Title: Immediate Effect of One-session Matrix Rhythm Therapy on the Functional Status and Treatment Satisfaction of Hemiparetic Patients
Brief Title: Immediate Effect of One-session MRT in Hemiparetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, PT.,PhD, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22.09.2021-MRT
Record Dates: First submitted 2021-09-22; First posted 2021-09-30 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hemiparesis;Poststroke/CVA; Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRT group (Experimental): One session Matrix-Rhythm Therapy
  Interventions: Other: Matrix-Rhythm Therapy
- Control group (Other): One session routine, conventional physiotherapy and rehabilitation
  Interventions: Other: Conventional physiotherapy and rehabilitation

INTERVENTIONS:
Other: Matrix-Rhythm Therapy — One session Matrix-Rhythm Therapy will be applied to affected body parts.
  Arms: MRT group
Other: Conventional physiotherapy and rehabilitation — Hemiparetics wil receive one session conventional physiotherapy and rehabilitation.
  Arms: Control group

SUMMARY:
Immediate effect of one-session Matrix Rhythm Therapy on the functional status and treatment satisfaction of hemiparetic patients will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* to have single-sided hemiparesis for the first time,
* to have hemiparesis at least four weeks earlier,
* to have Modified Rankin Score of ≤3

Exclusion Criteria:

* to use a cardiac pacemaker,
* to have communication problems,
* to have other neurological, psychiatric and/or orthopedic problems other than hemiparesis.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Motricity Motor Scale | 5 minutes
  Index for motor impairment after stroke
Trunk Impairment Scale | 10 minutes
  It consists of 3 subscales of static and dynamic sitting balance and trunk coordination
The Box and Block Test | 2 minutes
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
The Nine-Hole Peg Test | 2 minutes
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. Administered by asking the client to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible.
Treatment Satisfaction Scale | 30 sec.
  The amount of satisfaction that a patient feels ranges across a continuum from none (0) to an extreme amount of satisfaction (10).

SECONDARY OUTCOMES:
Global Rating of Change Scale | 30 sec.
  Global Rating of Change (GRC) scales provide a means of measuring self-perceived change in health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)